CLINICAL TRIAL: NCT04333719
Title: Prevalence of Deep Sedation in Terminal Palliative Phase
Acronym: PREVAL-S2P
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/02
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Palliative Care; Deep Sedations
Keywords: palliative care; prevalence; terminal phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- terminally ill patients in specialized palliative: terminally ill patients in specialized palliative care facilities
  Interventions: Other: Type of sedations

INTERVENTIONS:
Other: Type of sedations — Estimate the prevalence of deep sedations (i.e. with a -4 or -5 score at the Richmond scale at the induction time) for patients in terminal phase and receiving cares from a specialized palliative care facility

SUMMARY:
This nation-wide, multicentric, prospective and cross-sectional study aims to estimate the prevalence of deep sedations (i.e. with a -4 or -5 score at the Richmond scale at the induction time) for patients in terminal phase and receiving cares from a specialized palliative care facility (palliative care units, dedicated beds in acute units, mobile teams for inpatient or outpatients or home-based structures) in France.

DETAILED DESCRIPTION:
Inducing a deep sedation in palliative care is a sensitive practice. The abolition of the communication in a crucial moment of life for the patients is particularly challenging. This practice implies particular experiences for families and caregivers, often increased by the deepness of the sedation. In France, the Claeys-Leonetti law has added additional indications of deep sedation. The lack of data on the prevalence of this practice in palliative care complicates the implementation of research projects and the improvement of professionals skills. In existing literature, the proportions of patients thus sedated varied from 2.5 to 14.5%. To our knowledge, no study on the prevalence of deep sedative practices in terminal diseases has been carried out in France. This observational study will help to better understand the real importance of this practice among each palliative care structures. They will also serve to build research projects on this theme supporting improvement of care for this population.

In this study, the deep sedation is defined as a sedation directly inducing from the induction time a score of -4 or -5 at the Richmond vigilance scale (or a clinically equivalent state for the investigator) as defined by the French society of palliative care and accompanying.

The day of inclusion, the investigator will collect the information about the structure of palliative care (type, team composition, number of patients with an on-going terminal disease), the characteristics of the sedated patient(s) (age, disease, treatments) and of the sedation (sedative molecules, assessment of vigilance, consents and decision-making process). In case of an on-going sedation previously initiated but still in progress the day of inclusion, the investigator will retrospectively collect the required data.

ELIGIBILITY:
Inclusion Criteria:

* Major, minor, major with legal protection patient
* Follow-up by a specialized palliative care facility;
* Palliative situation of a disease (non-curable);
* In terminal palliative phase (life expectancy estimated by the investigator =< 4 weeks)

Exclusion Criteria:

* Not followed by a specialized palliative care facility;
* In curative situation (curable);
* In non-terminal palliative phase (life expectancy estimated by the investigator > 4 weeks).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Major, minor, major with legal protection patient, follow-up by a specialized palliative care facility, palliative situation of a disease (non-curable) in terminal palliative phase (life expectancy estimated by the investigator =< 4 weeks)
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Determine the number of patient with deep sedation | Day 1
  The primary endpoint will be the prevalence of deep sedations among all the included patients with a terminal disease receiving cares from a specialized palliative care facility.
Determine the number of patient with deep sedation | Day 31
  The primary endpoint will be the prevalence of deep sedations among all the included patients with a terminal disease receiving cares from a specialized palliative care facility.
Determine the number of patient with deep sedation | Month 60
  The primary endpoint will be the prevalence of deep sedations among all the included patients with a terminal disease receiving cares from a specialized palliative care facility.

SECONDARY OUTCOMES:
Determine the number of patient by type of disease | Day 1
  deep palliative sedations for each sub-group of duration, depth and consent regarding the SEDAPALL classification
Determine the number of patient by type of disease | Day 31
  deep palliative sedations for each sub-group of duration, depth and consent regarding the SEDAPALL classification
Determine the number of patient by type of disease | Day 60
  deep palliative sedations for each sub-group of duration, depth and consent regarding the SEDAPALL classification
Describe the sedative therapies used | Day 1
  Comparative of sedative therapies used
Describe the sedative therapies used | Day 31
  Comparative of sedative therapies used
Describe the sedative therapies used | Day 60
  Comparative of sedative therapies used

CONTACTS AND LOCATIONS:
Overall Officials: Benoît BURUCOA, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux - St André, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No